CLINICAL TRIAL: NCT07109115
Title: The Effects of Vitamin C on Exercise-Induced Oxidative Stress in Postmenopausal Females
Brief Title: The Effects of Vitamin C on Acute-Exercise in Postmenopausal Females
Acronym: PM-VitC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 302767
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Females; Males; Menopause; Sedentary; Healthy Participants
Keywords: Vitamin C; Postmenopausal Females; Exercise; Oxidative Stress; Vascular Health
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator 1: 200mg vitamin C (Experimental): Subjects will supplement with 200mg of vitamin C 2x a day for 3 days. 100mg will be taken in the morning and 100mg in the evening. On the 3rd day, subjects will be scheduled to return for post-supplementation testing and be instructed to take a full 200mg dose 30-minutes prior to arriving.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Active Comparator 1: 500mg vitamin C (Experimental): Subjects will supplement with 500mg of vitamin C 2x a day for 3 days. Subjects will take half the dose in the morning and half the dose in the evening. On the 3rd day, subjects will be scheduled to return for post-supplementation testing and be instructed to take a full dose 30-minutes prior to arriving.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Active Comparator 1: 1000mg vitamin C (Experimental): Subjects will supplement with 1000mg of vitamin C 2x a day for 3 days. Subjects will take half the dose in the morning and half the dose in the evening. On the 3rd day, subjects will be scheduled to return for post-supplementation testing and be instructed to take a full dose 30-minutes prior to arriving.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Placebo Comparator 1: 0mg Vitamin C (Placebo Comparator): Subjects will supplement with 0mg of vitamin C 2x a day for 3 days. Subjects will take half the dose in the morning and half the dose in the evening. On the 3rd day, subjects will be scheduled to return for post-supplementation testing and be instructed to take a full dose 30-minutes prior to arriving.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)

INTERVENTIONS:
Dietary Supplement: Vitamin C (Ascorbic Acid) — Subjects will be supplemented with the following vitamin C doses: 0mg, 200mg, 500mg, 1000mg.

SUMMARY:
This study is looking at whether vitamin C can help improve oxidative stress and blood vessel health in females after menopause. We will see if taking different amounts of vitamin C for a few days changes how the body handles stress from exercise. This could lead to safer ways to protect females from heart disease without using hormone therapy.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the leading cause of death in the United States. After menopause, females face a significantly increased risk of CVD due to declines in estrogen, which negatively impact nitric oxide (NO) production and vascular health. This coincides with an increase in reactive oxygen species (ROS), leading to an imbalance in redox signaling that may blunt beneficial adaptations to exercise.

Vitamin C (ascorbic acid) is a potent antioxidant that may restore redox balance and endothelial function. However, most studies have been conducted in males using high doses that may suppress beneficial ROS signaling. In contrast, this trial focuses on the dose-response effects of short-term vitamin C supplementation (200 mg, 500 mg, and 1000 mg/day for 3 days) on ROS/NO balance, both at rest and in response to acute exercise, in PMF versus age-matched males.

The study includes 15 sedentary PMF and 15 sedentary age-matched males, ages 45 and older. Participants complete 5-6 total study visits: one baseline/screening visit and four intervention visits in a randomized crossover design. Each intervention visit consists of 3 days of supplementation followed by fasting blood draws, vascular testing, and a 200-kcal high-intensity exercise bout on a cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal (for females; defined as no menstrual cycle for 1-year)
* Sedentary (<150min of moderate-intensity exercise per week or not engaged in a regular exercise program)
* Non-smoking
* Weight stable (+/-3 kg over the past 3 months)

Exclusion Criteria:

* Overt CVD
* Any condition or medication contraindicating safe exercise
* Hormone replacement therapy (last 3-months)
* Use of vasoactive medications (e.g., calcium channel blockers, statins, ACE inhibitors, ARBs, nitrates, alpha-/beta-blockers, diuretics), diabetes, or unstable medication regimens
* Diabetes
* Oral antibiotic use within previous four weeks
* Oral disease or poor oral health as determined by the Oral Health Questionnaire
* Using an antibacterial mouthwash or a mouthwash containing chlorhexidine and unwilling to discontinue use
* Cancer diagnosis

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Flow-Mediated Dilation (FMD%) - Brachial Artery Endothelial Function | 5x: Baseline/un-supplemented; after 3-days of 200mg of vitamin C supplementation; after 3-days of 500mg of vitamin C supplementation; after 3-days of 1000mg of vitamin C supplementation; after 3-days of 0mg of vitamin C/placebo supplementation
  Brachial artery endothelial function will be measured by flow-mediated dilation (FMD) in each participant 5x (at baseline and after 0mg (placebo) 200mg, 500mg, and 1000mg of vitamin C). Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation (250mmHg), and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle.
Basal ROS Concentrations - plasma 8-Isoprostane (8-iso) and malondialdehyde (MDA) | baseline and after 0mg/placebo, 200mg, 500mg, and 1000mg dose of vitamin C for 3-days each
  A venous blood sample will be collected from a vein in the antecubital fossa. Plasma will be separated out and stored at -80C until concentrations of 8-Isoprostane (8-iso) and malondialdehyde (MDA) are measured via commerically available ELISA kits. ROS concentrations will be measured at 5x points: at baseline and after 0mg (placebo), 200mg, 500mg, and 1000mg of vitamin C
Resting ROS/NO Balance - plasma N-oxides (nitrite and nitrate) | Baseline and after 3-days of placebo, 200mg, 500mg, and 1000mg doses of vitamin C
  Venous blood samples will be collected from an antecubital fossa vein. Plasma will be separated out and stored at -80C until analysis. Plasma N-oxides (nitrite and nitrate) will be evaluated from the plasma via ozone-based chemiluminescence using a Sievers NOA model 280i. The N-oxides will be compared with the basal ROS also measured to calculate a ROS/NO balance.
Exercise-Induced ROS (plasma 8-Isoprostane (8-iso) and malondialdehyde (MDA)) and NO (plasma nitrate and nitrite) | 16x points: 4 exercise session with blood will be collected immediately before, immediately after, 15-min after, and 30-min after exercise
  An intravenous catheter will be placed into a vein in the antecubital fossa. Participants will complete 4 high-intensity exercise sessions (~200kcals). Each exercise session will be after 3-days of vitamin C supplementation (0mg/placebo, 200mg, 500mg, and 1000mg). Blood will be collected immediately before, immediately after, 15-min after, and 30-min after exercise. Plasma will be separated out and used to evaluate the changes in ROS (plasma 8-Isoprostane (8-iso) and malondialdehyde (MDA)) and NO (plasma nitrate and nitrite) from baseline/rest.

SECONDARY OUTCOMES:
Vitamin C | 5x points over 5-6 weeks: (1) baseline/unsupplemented and after 3-days of (2) 0mg/placebo, (3) 200mg, (4) 500mg, and (5) 1000mg of vitamin C supplementation
  Blood samples will be collected to evaluate compliance. We will measure vitamin C concentrations after each supplementation phase.
Oral Nitrate Reducing Capacity | 5x points over 5-6 weeks: (1) baseline/unsupplemented and after 3-days of (2) 0mg/placebo, (3) 200mg, (4) 500mg, and (5) 1000mg of vitamin C supplementation
  Assessment of the oral microbiome's ability to reduce nitrate to nitrite. This will be measured through an unstimulated saliva sample and a rinse of a standard nitrate solution.
Pulse Wave Analysis and Velocity | 5x points over 5-6 weeks: (1) baseline/unsupplemented and after 3-days of (2) 0mg/placebo, (3) 200mg, (4) 500mg, and (5) 1000mg of vitamin C supplementation
  Brachial artery blood pressures will be obtained using a standard sphygmomanometer. Aortic blood pressures will be obtained using applanation tonometry (SphygmoCor version 8.0, AtCor Medical).
Microvascular Function | 5x points over 5-6 weeks: (1) baseline/unsupplemented and after 3-days of (2) 0mg/placebo, (3) 200mg, (4) 500mg, and (5) 1000mg of vitamin C supplementation
  Participants will remain in a supine position with their left or right forearm slight extended and supinated. The cuff used for FMD will remain in place and two circular discs will be placed on the participants extended forearm. A laser Doppler imager (Moor Instruments - FLPI2) will be positioned directly over the participants forearm to measure skin blood flow in three different ways: microvascular flow mediated dilation, acetylcholine, and local thermal heating.
Exercise Capacity | Baseline only
  Participants will exercise using an incremental cycle ergometer protocol with increasing power output until volitional exhaustion is reached. The power output will increase in 3-minute stages, where blood is collected before the start of exercise and at the end of each stage. The LT will be established by analyzing the blood lactate-power output relationship. VO2 peak will be defined as the highest one min value attained during the test.
Tissue Perfusion (NIRS) | 5x points over 5-6 weeks: (1) baseline/unsupplemented and after 3-days of (2) 0mg/placebo, (3) 200mg, (4) 500mg, and (5) 1000mg of vitamin C supplementation
  Tissue oxygenation will be captured noninvasively using non-invasive, near-infrared spectrometry (NIRS, PortaMon, Artinis Medical Systems B.V., The Netherlands) positioned on the gastrocnemius (calf) or vastus lateralis (quad) muscle during the VO2/LT test and during each Experimental Visit (HIE sessions).
Central Hemodynamics (Physioflow) | 5x points over 5-6 weeks: (1) baseline/unsupplemented and after 3-days of (2) 0mg/placebo, (3) 200mg, (4) 500mg, and (5) 1000mg of vitamin C supplementation
  : Measures of central hemodynamics (cardiac output, etc.) will be non-invasively captured throughout the VO2/LT test and during each Experimental Visit (HIE sessions). Using electrodes placed on the participant's body and the principles of signal morphology impedance cardiography PhysioFlow provides estimates of central cardiac measures at rest and during exercise non-invasively.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, PhD, Principal Investigator — UVA

IPD SHARING:
Plan to Share IPD: No